CLINICAL TRIAL: NCT05286840
Title: 64Cu-SAR-bisPSMA Positron Emission Tomography of Patients With Known or Suspected Prostate Cancer: A Prospective, Non-randomized, Single Arm, Single Center, Open-label Phase 1/2 Study
Brief Title: 64Cu-SAR-bisPSMA Positron Emission Tomography of Patients With Known or Suspected Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Luke Nordquist, MD (Other)
Collaborators: Clarity Pharmaceuticals (Unknown)
Responsible Party: Sponsor-Investigator, Luke Nordquist, MD, Sponsor/Principal Investigator, GU Research Network, LLC
Organization: GU Research Network, LLC (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GU22-002
Record Dates: First submitted 2022-02-28; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective, non-randomized, single arm, single center, open-label study .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 64Cu-SAR-bisPSMA — Diagnostic PET/CT imaging agent targeted for Prostate Specific Membrane Antigen (PSMA)

SUMMARY:
This research project is testing a new compound which may potentially detect specific cancer lesions in men with prostate cancer.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single arm, single center, open-label study of 64Cu-SAR-bisPSMA PET in patients with known or suspected prostate cancer (PC).

Patients will be screened during a 28-day period and assessed against the inclusion and exclusion criteria. During screening the investigator will determine the patient's disease status (for patients with suspected prostate cancer) or stage of disease (for patients with known prostate cancer) and management plan based on the available standard of care test results (including available imaging, histopathology, biochemical markers, clinical and symptoms history, etc.). Eligible patients will receive a single administration of 64Cu-SAR-bisPSMA and complete a PET scan at an early time (1-4 hours) and a late time (24-72 hours).

The patient's status will only be assessed in patients with suspected disease at study entry and will be characterized as suspected or known prostate cancer during the follow up.

Staging will only be assessed in patients with known prostate cancer at study entry and will be characterized according to the TNM system and as Localized, Regional or Distant (nodes/visceral/bone).

ELIGIBILITY:
Inclusion Criteria:

1. Signed an informed consent.
2. >18 years of age.
3. Known diagnosis of prostate adenocarcinoma confirmed by histopathology OR patients with suspicion of prostate cancer based on elevated PSA but negative standard of care imaging and/or negative biopsy.
4. The Eastern Cooperative Oncology (ECOG) performance status 0-2.
5. Adequate recovery from acute toxic effects of any prior therapy.
6. Adequate renal function (eGFR of 30 ml/min/1.73m2 or higher)

Exclusion Criteria:

1. Participants must not receive other investigational agents within 28 days prior to 64Cu-SAR-bisPSMA administration.
2. Patients administered any high energy (>300 KeV) gamma-emitting radioisotope within 5 physical half-lives prior to 64Cu-SAR-bisPSMA administration.
3. Known or expected hypersensitivity to 64Cu-SAR-bisPSMA or any of its components.
4. Any serious medical condition or extenuating circumstance which the investigator feels may interfere with the procedures or evaluations of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2022-03-28 (Estimated); Primary Completion 2023-03-28 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
To assess safety of 64Cu-SAR-bisPSMA (all patients). | From injection of 64Cu-SAR-bisPSMA to one week following.
  To assess treatment emergent adverse events.

SECONDARY OUTCOMES:
Disease status adjustment (patients with suspected disease at entry) before vs after 64Cu-SAR-bisPSMA PET/CT Imaging. | Within one week of 64Cu-SAR-bisPSMA PET/CT Imaging
  Disease status will be assessed before and after 64Cu-SAR-bisPSMA PET/CT Imaging.
Disease Staging adjustment (for patients with known disease at entry) before vs after 64Cu-SAR-bisPSMA PET/CT Imaging. | Within one week of 64Cu-SAR-bisPSMA PET/CT Imaging
  Disease staging will be assessed before and after 64Cu-SAR-bisPSMA PET/CT Imaging
Clinical Management plan before vs after 64Cu-SAR-bisPSMA PET/CT Imaging. | Within one week of 64Cu-SAR-bisPSMA PET/CT Imaging
  Clinical Management plan will be documented before and after 64Cu-SAR-bisPSMA PET/CT Imaging.

OTHER OUTCOMES:
Disease detection ability of 64Cu-SAR-bisPSMA PET (all patients). | Within one week of 64Cu-SAR-bisPSMA PET/CT Imaging
  64Cu-SAR-bisPSMA PET/CT Imaging will be used to detect prostate cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- GU Research Network, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No